CLINICAL TRIAL: NCT00125424
Title: A Randomized, Double-Blind, Dose-Response Study to Assess the Efficacy and Safety of AQUAVAN® Injection for Procedural Sedation in Patients Undergoing Colonoscopy
Brief Title: Study of AQUAVAN® Injection (AQUAVAN; Fospropofol Disodium) for Sedation During Colonoscopy
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 3000-0520; GPI 3000-0520
Record Dates: First submitted 2005-07-27; First posted 2005-08-01 (Estimated); Last update posted 2008-11-07 (Estimated); Status verified 2008-11

CONDITIONS: Colonoscopy; Colonic Polyps
Keywords: Colonoscopy; Sedation; AQUAVAN; (fospropofol disodium); Endoscopic sedation; Endoscopic outcomes; Endoscopy
MeSH Terms: conditions — Colonic Polyps | interventions — fospropofol; Injections; Midazolam

INTERVENTIONS:
Drug: AQUAVAN® (fospropofol disodium) Injection
Drug: Midazolam HCl

SUMMARY:
Very often, patients receive sedative medication before a diagnostic, therapeutic, or surgical procedure to help them relax, keep them calm, and to relieve them from pain. This is called procedural sedation. During procedural (mild to moderate) sedation, a patient is first given a pain-relief medication (analgesic) and then a medication to help him/her relax and keep him/her calm (sedative). Propofol is the drug commonly used for sedation because it releases immediately into the blood stream and causes fast sedation. AQUAVAN (fospropofol disodium) is made as a slow release version of propofol, allowing for fast sedation and possibly faster recovery and discharge.

This study is intended to compare several different doses of AQUAVAN in patients having a colonoscopy in order to find the right dose that will get patients to a level of mild to moderate (procedural) sedation.

DETAILED DESCRIPTION:
This is a randomized, double-blind study designed to evaluate the dose-response in the sedation success rate for 4 different initial bolus doses of AQUAVAN following pretreatment with an analgesic, fentanyl, in patients undergoing a colonoscopy. A group of patients will receive midazolam as a reference therapy.

Following completion of pre-procedure assessments, patients will be randomly assigned to 1 of 5 IV treatment groups at an equal allocation ratio (25 patients per arm) on the day of the scheduled procedure. Randomization will be stratified by age and ASA status:

AQUAVAN initial bolus dose 1: 8 mg/kg AQUAVAN initial bolus dose 2: 6.5 mg/kg AQUAVAN initial bolus dose 3: 5 mg/kg AQUAVAN initial bolus dose 4: 2 mg/kg Midazolam initial bolus dose: 0.02 mg/kg

A person skilled in airway management and authorized by the facility in which the colonoscopy is performed (such as a respiratory therapist, a study nurse, or a clinician) must be immediately available during the conduct of the study. All patients will be placed on supplemental oxygen via nasal cannula (4 L/min), and a 12-lead electrocardiogram (ECG), pulse oximeter, and blood pressure monitor prior to administration of study medication. All patients will receive an injection of analgesic pretreatment followed by the administration of sedative medication, as described below. This protocol recognizes 2 distinct phases of sedation: Sedation Initiation and Sedation Maintenance. Assessments will be made to evaluate the patients for levels of sedation, clinical benefit, and adverse events as detailed in the protocol. Blood samples will be collected for pharmacokinetic (PK) analysis, also detailed in the protocol.

ELIGIBILITY:
- Number of Patients/Site: Approximately 125 patients, 25 per arm, at up to 25 sites will be randomized into this study.

- Study Country Location: United States

- Study Population: Male and female patients aged 18 years and older and undergoing elective colonoscopy will be enrolled in the study.

Inclusion Criteria:

1. Patient provides signed/dated informed consent and Health Insurance Portability and Accountability Act of 1996 (HIPAA) authorization after receiving a full explanation of the extent and nature of the study
2. Patient must be at least 18 years of age at the time of screening
3. If female, patient must be surgically sterile, postmenopausal, or not pregnant or lactating and has been using an acceptable method of birth control for at least 1 month prior to dosing, with a negative urine pregnancy test result at screening and pre-dose
4. Patient meets American Society of Anesthesiologists (ASA) Physical Classification System status of P1 to P4

Exclusion Criteria:

1. Patient has a history of allergic reaction or hypersensitivity to any anesthetic agent, narcotic, or benzodiazepine
2. Patient does not meet nils per os (NPO) status per ASA guidelines or institution's guidelines
3. Patient has a Mallampati classification score of 4; OR a Mallampati classification score of 3 AND a thyromental distance <= 4 cm, or for any other reason has a difficult airway, in the opinion of the Investigator
4. Patient has an abnormal, clinically significant 12-lead ECG finding at predosing period Day 0
5. Patient has participated in an investigational drug study within 1 month prior to study start
6. Patient is unwilling to adhere to pre- and post-procedural instructions
7. Patient for whom the use of fentanyl is contraindicated
8. Patient for whom the use of Midazolam HCl injection (Midazolam) is contraindicated

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125
Dates: Start 2005-07; Study Completion 2005-09 (Actual)

PRIMARY OUTCOMES:
Three consecutive MOAA/S scores ≤4 after administration of sedative medication AND completing the procedure without requiring the use of alternative sedative medication AND without requiring manual or mechanical ventilation

SECONDARY OUTCOMES:
Patient's rating of experience after ready for discharge
Principal Investigator's (PI's) rating at end of procedure
Percentage of patients requiring alternative sedative medication
Number of doses/amount of fentanyl administered
Number of doses of study medication administered
Time to sedation, digital rectal examination, start of procedure, reach splenic flexure, hepatic flexure, cecum, end of procedure, and ready for discharge
Percentage of patients requiring repositioning
Percentage of patients whose procedures are interrupted due to inadequate sedation
Time to ready for discharge from end of procedure
Change from baseline DSST score over time during recovery period
Patient's rating at 24 hour post discharge telephone survey
Duration and percent of time when a patient's MOAA/S score is at each level between the first dose of study medications and fully alert and during the procedure
PI's rating of level of sedation prior to initiation of the procedure
Percentage of patients with a mean MOAA/S of 2 to 4 and 0 to 1 during the procedure
MOAA/S over time

CONTACTS AND LOCATIONS:
Overall Officials: James Jones, PharmD, MD, Study Director — Eisai Inc.
Locations (20):
- United States (20):
  - Clinical Research Associates, Huntsville, Alabama
  - Arizona Research Center, Phoenix, Arizona
  - Atlanta Gastroenterology Associates, Atlanta, Georgia
  - Rockford Gastroenterology Associates Ltd., Rockford, Illinois
  - Welborn Clinic, Evansville, Indiana
  - Gulf Coast Research Associates, Inc., Baton Rouge, Louisiana
  - Gastroenterology Clinic, Monroe, Louisiana
  - Chevy Chase Clinical Research, Chevy Chase, Maryland
  - Endoscopic Microsurgery Associates, PA, Towson, Maryland
  - Gastrointestinal Associates, PA, Jackson, Mississippi
  - Winthrop-University Hospital, Mineola, New York
  - Research Associates of New York, New York, New York
  - Asheville Gastroenterology Associates/The Endoscopy Center, Asheville, North Carolina
  - Oklahoma Gastroenterology Associates, Tulsa, Oklahoma
  - Memphis Gastroenterology Group, PC, Memphis, Tennessee
  - Gastrointestinal Institute, Nashville, Tennessee
  - St. Thomas Medical Group, P.C., Nashville, Tennessee
  - Alamo Research Center, San Antonio, Texas
  - Spokane Digestive Diseases Center, Spokane, Washington
  - Wisconsin Center for Advance Research, Milwaukee, Wisconsin